CLINICAL TRIAL: NCT00501319
Title: Longitudinal Measurement of Pain and Other Symptoms of Non-Small Cell Lung Cancer (NSCLC) Patients Following Thoracic Surgery
Brief Title: Measurement of Pain and Other Symptoms of Non-Small Cell Lung Cancer (NSCLC) Patients Following Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: ID02-320
Record Dates: First submitted 2007-07-12; First posted 2007-07-16 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Lung Cancer
Keywords: Interactive Voice Response Telephone System; Non-Small Cell Lung Cancer; Lung Cancer; Questionnaire; Survey; NSCLC; IVR
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Non-Small Cell Lung Cancer.
  Interventions: Behavioral: Interactive Voice Response (IVR); Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Interactive Voice Response (IVR) — Phone calls once weekly for the first 3 months after surgery, then every two weeks for an additional 3 months.
Behavioral: Questionnaire — Questionnaires taking 20 minutes to complete.
  Other Names: Survey

SUMMARY:
Primary Objectives:

* To longitudinally assess the natural history of symptoms (prevalence, severity, patterns of symptoms, and the relationship of physical and psychological distress) among post-thoracic surgery for non-small cell lung cancer patients with early stage (stage I-IIIA) disease.
* To determine crisis events (when symptoms are most severe), their relationship with cancer therapy, surgical techniques and disease, and their relationship with function and quality of life; and to determine current practice patterns of symptom control throughout the six months of the post-surgical phase.
* To determine the utility of a weekly, telephone-administered interactive voice response symptom assessment (IVR-MDASI) for identifying emergent clinically significant symptoms in this population.
* To develop symptom severity critical values and critical treatment algorithms for post-operative symptom control for NSCLC patients.

DETAILED DESCRIPTION:
Before surgery, you will be asked to complete four surveys about your mood, symptoms, quality of life, and smoking history. Completing the questionnaires will take about 20 minutes. You will be asked for some information about age, sex, race, education, marital status, and employment status (full-time, part-time, unemployed). Before surgery, the research nurse will teach you how to use the special telephone system, called an Interactive Voice Response (IVR) telephone system. This system is used for tracking symptoms at home. An instruction pamphlet will also be given to you.

Three days after surgery, while you are in the hospital, you will be asked by the research nurse to again complete one questionnaires that measures your symptoms.

Once you are home from the hospital, the automatic telephone IVR system will call at a prescheduled time that is convenient for you. The phone call will take about four minutes to complete. The IVR will call once a week for the first 3 months after surgery, and then every two weeks for an additional 3 months.

The research nurse will call you one week after surgery and then one month, three months, and six months to complete four questionnaires about symptoms, mood, quality of life, and smoking history. It will take about 20 minutes to complete the questionnaires.

The information collected by the IVR is for research purposes only, and you must report any symptoms that you are concerned about to your physicians or nurses.

Should severe symptoms develop, research staff will notify the your treatment team.

This is an investigational study. About 112 patients will participate in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for thoracic surgery for NSCLC (stage I-IIIA)
* Patients >/= 16 years of age
* Patients who speak English
* Patients residing in the United States

Exclusion Criteria:

* Current diagnosis of psychosis or dementia
* Patients who have difficulty understanding the intent of the study
* Patients who can not complete the assessment tools
* Patients without telephone access

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Non-Small Cell Lung Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2003-04; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To study the symptoms of patients who receive thoracic surgery for the treatment of lung cancer. | 6 Years

SECONDARY OUTCOMES:
To test the usefulness of a special telephone system for tracking the symptoms of patients after they have had thoracic surgery. | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Xin Shelley Wang, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org